CLINICAL TRIAL: NCT06721286
Title: Toripalimab Combined With Gemcitabine and Cisplatin (GemCis) as Preoperative Neoadjuvant Therapy for Resectable Intrahepatic Cholangiocarcinoma (ICC) With High Risk of Recurrence, Phase II, Single-center, Randomized Controlled Trial
Brief Title: Toripalimab Combined With Gemcitabine and Cisplatin (GemCis) as Preoperative Neoadjuvant Therapy for Resectable Intrahepatic Cholangiocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20241190
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: Intrahepatic Cholangiocarcinoma (Icc)
Keywords: Intrahepatic Cholangiocarcinoma; neoadjuvant therapy; toripalimab
MeSH Terms: conditions — Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension | interventions — Gemcitabine; Cisplatin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative neoadjuvant therapy group (Experimental)
  Interventions: Drug: Teripalimab; Drug: Gemcitabine + Cisplatin; Procedure: Surgery
- Control group (Experimental)
  Interventions: Procedure: Surgery

INTERVENTIONS:
Drug: Teripalimab — 240mg intravenous injection, D1, q3w, for 9 weeks (3 cycles)
  Arms: Preoperative neoadjuvant therapy group
Drug: Gemcitabine + Cisplatin — Gemcitabine 1000mg/m2 + cisplatin 25mg/m2, D1&D8, q3w, for 9 weeks (3 cycles)
  Arms: Preoperative neoadjuvant therapy group
Procedure: Surgery — Radical resection

SUMMARY:
This study was a randomized controlled trial to evaluate the efficacy and safety of toripalimab combined with GemCis (gemcitabine and cisplatin) as preoperative neoadjuvant therapy for resectable ICC at high risk of recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18, male or female;
2. Pathological diagnosis confirmed intrahepatic cholangiocarcinoma, which could be resected surgically; One of the following conditions shall be met:

   2.1 Single tumor, diameter greater than 5cm (T1b) 2.2 Single tumor with vascular invasion (T2), multiple tumors ≤ 3 2.3 Tumor penetrating visceral peritoneum (T3) or directly invading surrounding organs (T4) 2.4 Suspicious lymph node metastasis in Zone 8, 12 or 13
3. Can not received systemic treatment before participating in the study;
4. ECOG PS score 0-1;
5. The main organs function normally, and there is no serious blood, heart, lung, liver, kidney, bone marrow and other functional abnormalities and immune deficiency diseases.
6. Laboratory inspection shall meet the following requirements:

   Women of childbearing age must have a negative pregnancy test (serum or urine) within 14 days before enrollment, and voluntarily use appropriate methods of contraception during the observation period and within 8 weeks after the last administration of the study drug; For men, they should be surgically sterilized or agree to use appropriate methods of contraception during the observation period and within 8 weeks after the last administration of the study drug.
7. The patient voluntarily participated and signed the informed consent form;
8. It is expected that the compliance is good, and the efficacy and adverse reactions can be followed up according to the requirements of the scheme.

Exclusion Criteria:

1. Patients who received PD-1, PD-L1, PD-L2, CTLA-4 before enrollment, or directly received another stimulatory or co inhibitory T cell receptor (such as CTLA-4, 0X40, CD137);
2. Any other research drugs within 4 weeks before enrollment;
3. Any active autoimmune disease or history of autoimmune disease (such as interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism after hormone replacement therapy);
4. Congenital or acquired immune function defects, such as human immunodeficiency virus (HIV) infection;
5. Uncontrollable clinical cardiac symptoms or diseases, such as NYHA II and above heart failure unstable angina pectoris, myocardial infarction within one year, and clinically significant supraventricular or ventricular arrhythmia requiring clinical intervention;
6. Severe infection (such as intravenous drip of antibiotics, antifungal or antiviral drugs) occurred within 4 weeks before the first drug administration, or fever of unknown cause>38.5 ° C occurred during screening/before the first drug administration;
7. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
8. Live attenuated vaccine shall be inoculated within 4 weeks before the first administration or planned during the study period;
9. Suffered from or accompanied by other system malignant tumors in the last 5 years (except cured skin basal cell carcinoma, cervical carcinoma in situ and ovarian cancer);
10. Allergic to any test drug;
11. Pregnant and lactating women, fertile subjects are unwilling to take effective contraceptive measures;
12. Uncontrollable psychosis;
13. Other situations that the researcher thinks are not suitable for inclusion. If the patient has central nervous system metastasis, has serious laboratory examination abnormalities, and is accompanied by family or social factors, it will affect the safety of the subject, or the collection of data and samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year recurrence-free survival rate | 1 year

SECONDARY OUTCOMES:
1-year OS | 1 year
2-year OS | 2-year
ORR | 1 year
DCR | 1 year
R0 resection rate | 1 year
30 day postoperative complication rate | 1 year
Occurrence of adverse reactions | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China